CLINICAL TRIAL: NCT02125864
Title: Plasma Levels of Vascular Endothelial Growth Factor Before and After Intravitreal Injection of Aflibercept in Patients With Exudative Age-related Macular Degeneration
Brief Title: Plasma Levels of Vascular Endothelial Growth Factor Before and After Intravitreal Injection of Aflibercept
Acronym: Eylea-2014
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, ANCA ROALD, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-000103-27
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: AMD; VEGF; Aflibercept
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept (Experimental): There is only one arm. Plasma VEGF is investigated in the same patient before and after intravitreal Aflibercept injection.
  Interventions: Procedure: intravitreal injection

INTERVENTIONS:
Procedure: intravitreal injection — collecting blood samples

SUMMARY:
The purpose of this study is to examine the plasma concentration of vascular endothelial growth factor (VEGF) after standard treatment with one of the newest growth factor inhibitors, aflibercept (Eylea).

Patients with exudative age-related macular degeneration (AMD) are treated today with anti-growth factors (anti-VEGF). Eylea appears to have a longer duration of action in the eye and a more powerful effect on the edema in the macula than previously used growth factor inhibitors. This means that the disease can be controlled with fewer number of injections into the eye and the investigators can therefore reduce the risk of complications associated with this type of treatment.

It is unclear what the plasma VEGF concentration after treatment with Eylea into the eye in patients with wet age-related macular degeneration is.

DETAILED DESCRIPTION:
Macular edema secondary to exudative age-related macular degeneration is treated today primarily with vascular endothelial growth factor inhibitors, anti-VEGF.

There are currently four anti-VEGF drugs that are either approved or off-label used in ophthalmology. Pegaptanib (Macugen, Pfizer), ranibizumab (Lucentis, Novartis) aflibercept (Eylea, Bayer) and bevacizumab Avastin, Roche) . They have different molecules and pharmacodynamics .

VEGF plays an important role in many physiological and pathophysiological mechanisms. Studies have shown that even low-dose intravitreal treatment with bevacizumab leads to significant reduction of VEGF plasma concentration up to a month after treatment in patients with exudative AMD.

No significant systemic effect could be detected after intravitreal administration of ranibizumab or pegaptanib.

The purpose of this study is :

* To determine if intravitreal treatment with Eylea affects VEGF plasma levels in patients with exudative AMD
* How long after intravitreal injection is VEGF plasma concentration affected?

ELIGIBILITY:
Inclusion Criteria:

* Men and women with exudative AMD
* Central Retinal Thickness ≥ 250 microns
* Best corrected visual acuity 20/25-20/320
* Age ≥ 60 years
* Only one eye will be applicable for recruitment
* Informed signed consent according to International Conference on Harmonisation Good Clinical Practice should be in place prior to study .

Exclusion Criteria:

* Bilateral disease
* Treatment with intravitreal injections in the past three months
* Patients who have previously undergone vitrectomy
* Choroidal neovascular membrane secondary to other disease than AMD
* Macula edema of other etiology than wet AMD
* Intraocular pressure ≥ 30 mmHg in mydriasis
* Active uveitis or infectious condition in the study eye
* Patients using systemic anti inflammatory therapy ( steroids)
* Patients using systemic anti-VEGF treatment
* Blod pressure which is not well regulated
* Dialysis or in need of transplantation resulting from renal failure
* Heart attack, stroke, transient ischemic attack in the last 6 months
* New York Heart Association class II , III , IV
* Known allergy to aflibercept , fluorescein or povidone iodine
* Unable to follow the study procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mean change in VEGF plasma concentration (pg/mL) | 6 months

SECONDARY OUTCOMES:
Mean change in Visual Acuity as measured with the Snellen chart | 6 months
Central Retinal Thickness as measured by Optical coherence tomography expressed in microns | 6 months
Number of non-responders | 6 months

REFERENCES:
- [Derived] Roald AB, Aass HC, Moe MC. Recovery of plasma vascular endothelial growth factor concentrations during aflibercept loading phase and after the transition to bimonthly treatment for neovascular age-related macular degeneration. Br J Ophthalmol. 2015 Dec;99(12):1610-3. doi: 10.1136/bjophthalmol-2015-306781. Epub 2015 May 12. PMID 25966740